CLINICAL TRIAL: NCT04917276
Title: Treatment Response Prediction System of Metastatic Colorectal Cancer Based on Circulating Tumor Cells
Brief Title: Treatment Response Prediction System of mCRC Patients Based on CTC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: ZSCTC2
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-04

CONDITIONS: Colorectal Cancer Stage IV; Circulating Tumor Cell
MeSH Terms: conditions — Colorectal Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training Group: The training cohort that used to built the response prediction model
  Interventions: Diagnostic Test: Circulating tumor cell
- Validation Group: The validation cohort that used to validate the response prediction model
  Interventions: Diagnostic Test: Circulating tumor cell

INTERVENTIONS:
Diagnostic Test: Circulating tumor cell — Detecting CTC in different time points of treatment (like PR, PD, pre and post-operation)

SUMMARY:
This study enrolling patients with metastatic colorectal cancer. Detecting CTC at different points in the treatment process. Descripting the molecular atlas of CTC in mCRC patients. Building and validating a response prediction system of mCTC patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years;

histologically proven colorectal liver metastasis

With liver-dominant disease (extrahepatic metastases limited to lung metastases)

ECOG 0-1

A life expectancy of ≥ 3 months

Adequate hematologic function: absolute neutrophil count (ANC)≥1.5×109/l, platelets≥75×109/l, and international normalized ratio (INR) ≤1.3

Adequate liver and renal function: total bilirubin ≤2.0 mg/dl, alanine aminotransferase, aspartate aminotransferase ≤ 5x upper limit of normal, and albumin≥2.5 g/dl, serum creatinine≤2.0 mg/dl

Written informed consent for participation in the trial.

Exclusion Criteria:

* Other previous malignancy within 5 years

Have metastases other than liver and lung metastases

Receiving any treatment before first blood collection

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer (with lung or liver metastases) who receiving chemotherapy with or without target therapy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 1 year
  The sensitivity of the response prediction model
Specificity | 1 year
  The specificity of the response prediction model

IPD SHARING:
Plan to Share IPD: Undecided